CLINICAL TRIAL: NCT03808987
Title: TRANSFORM: Translational Research That Adapts New Science FOR Maltreatment Prevention
Brief Title: Promotion of Successful Parenting
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sheree Toth, Director, Mt. Hope Family Center, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1P50HD096698-01 (NIH); 1P50HD096698-01 (NIH)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-04

CONDITIONS: Pregnant and Parenting Women
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Child-Parent Psychotherapy
Who Masked: Outcomes Assessor
Masking Description: Research assistants will be blind to the arm the participant has been randomly assigned to and to study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CHW+CPP brief prenatal onset (Experimental): Participants will receive Child-Parent Psychotherapy (CPP) for 6 months, beginning prenatally, in addition to services from a Community Health Worker (CHW)
  Interventions: Behavioral: Child-Parent Psychotherapy (CPP); Behavioral: Community Health Worker (CHW) home visitation
- CHW+CPP brief postnatal onset (Experimental): Participants will receive Child-Parent Psychotherapy (CPP) for 6 months, beginning postnatally, in addition to services from a Community Health Worker (CHW)
  Interventions: Behavioral: Child-Parent Psychotherapy (CPP); Behavioral: Community Health Worker (CHW) home visitation
- CHW+CPP 12 months (Experimental): Participants will receive Child-Parent Psychotherapy (CPP) for 12 months, beginning prenatally, in addition to services from a Community Health Worker (CHW)
  Interventions: Behavioral: Child-Parent Psychotherapy (CPP); Behavioral: Community Health Worker (CHW) home visitation
- CHW only (Experimental): Participants will receive services from a Community Health Worker (CHW) without Child-Parent Psychotherapy (CPP)
  Interventions: Behavioral: Community Health Worker (CHW) home visitation

INTERVENTIONS:
Behavioral: Child-Parent Psychotherapy (CPP) — Child-Parent Psychotherapy (CPP) focuses on parent-infant relationships, increases efficacy for improved mother-child relationships, more sensitive parenting, healthier child development, and maltreatment prevention. A primary goal is to strengthen the parent-child relationship to improve family functioning and child security of attachment. Through respect, empathic concern, and positive regard, the therapeutic relationship provides mothers with corrective emotional experiences, through which they are able to differentiate current from past relationships, form positive internal representations of themselves and of themselves in relationship to others, particularly their children. Parents are encouraged to process their experiences of trauma and restore parental roles as protective shields, improve affective regulation capacities, enhance understanding of the meaning of behavior, acknowledge the impact of trauma, and support children in a more positive developmental trajectory.
  Arms: CHW+CPP 12 months; CHW+CPP brief postnatal onset; CHW+CPP brief prenatal onset
Behavioral: Community Health Worker (CHW) home visitation — Community Health Worker (CHW) home visitation includes assistance with concrete support needs, such as transportation to medical appointments, referrals for food, housing, and employment services, and attention to developmental needs of young children.

SUMMARY:
Home visitation by community health workers is a commonly utilized approach to support families and prevent child maltreatment. At times, however, more intensive intervention is needed to address familial trauma, depression, or other challenges. This preventive treatment evaluation study evaluates whether adding Child-Parent Psychotherapy (CPP) to a Community Health Worker (CHW) outreach model improves positive parenting and parent-child relationships above CHW alone. The efficacy of CPP has been demonstrated with maltreated and other high-risk populations. This evaluation will examine optimal timing of CPP (beginning prenatally or postnatally) and optimal duration of services (6 vs. 12 months). Additionally, how and for whom CPP is most effective and why will be examined. Assessments of parenting, maternal sensitivity, representational models, cognitions, physiological reactivity, and physical health indicators will be assessed prenatally, and at children's age of 3, 9, and 12 months.

DETAILED DESCRIPTION:
PROMISE is integrated into the TRANSFORM Capstone Center to promote the next generation of research on child maltreatment, translate research findings into clinical and preventive interventions, and disseminate research and best practice to varied stakeholders. Informed by developmental psychopathology, the research incorporates multiple levels of analysis within a lifespan framework. Increasing knowledge of optimal methods for delivering dual mother and child preventive intervention has crucial public health significance in preventing child maltreatment. PROMISE involves a randomized control trial to evaluate whether expanding a Community Health Worker (CHW) outreach model, by adding Child-Parent Psychotherapy (CPP), an intensive intervention that focuses on parent-infant relationships for families at risk for child maltreatment, increases efficacy for improved mother-child relationships, more sensitive parenting, healthier child development, and maltreatment prevention. The efficacy of CPP has been demonstrated with maltreated and other high-risk populations. Through the use of four intervention arms, the evaluation will assess whether more intensive intervention better protects against child maltreatment compared with CHW support alone, and will determine the optimal timing of these interventions (i.e., beginning prenatally or postnatally), the optimal duration of services (i.e., 6 vs. 12 months), mechanisms of effect (mediator analyses), and which intervention strategy works best for mothers with varying risk factors (moderator analyses). Pregnant women (N = 300) and their infants after birth will participate. Longitudinal assessments will occur during the third trimester of pregnancy, at infant's ages of 3 and 9 months, and a post-intervention follow-up at 15 months old. The measurements obtained at each timepoint constitute a rich multi-level perspective of maternal and child functioning over time in response to the interventions. Maternal parenting behaviors, representational models, cognitions, and physiological reactivity, and infants' health and development will be assessed longitudinally. CPP groups are hypothesized to improve sensitive and responsive parenting and secure attachment, relative to CHW home visitation alone, thereby reducing risks for child maltreatment. Improvements in maternal attachment representations, parenting cognitions, and stress reactivity are hypothesized to mediate treatment outcomes. Moderators, including maternal histories of trauma, psychopathology, and intimate partner violence, will advance determination of differential responsiveness to CHW and CPP (what works for whom and why?) and allow for tailored preventive strategies. Identification of timing, dosage, and intensity of service delivery, along with outcome mediators and moderators is innovative and will facilitate development of targeted prevention and intervention strategies that support parenting and decrease child maltreatment for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be low-income pregnant adult women eligible for Medicaid and who have been referred to a Community Health Worker program based on their high psychosocial risk status.

Exclusion Criteria:

* Mothers will be excluded if they have significant cognitive limitations, severe psychiatric disorders requiring a higher level of care (e.g., imminent suicidal ideation requiring hospitalization, psychotic features), non-English proficiency, age less than 18, or a physical disability that impedes ability to complete study procedures. Mothers whose psychiatric needs or substance use requires inpatient treatment will be excluded. Mothers will be excluded if they terminate their pregnancy or do not deliver a live birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrollment will include pregnant women
Enrollment: 222 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parental Sensitivity (measured with the Parental Bonding Questionnaire) | Assessment at child's age of 9 months
  Improvements in maternal reports of positive emotional responses to their babies
Parental Acceptance (measured with the Parental Acceptance and Rejection Questionnaire) | Assessment at child's age of 9 months
  Improvements in maternal reports of acceptance in parent-child relationships

SECONDARY OUTCOMES:
Parental Sensitivity (measured with the Parental Bonding Questionnaire) | Assessment at child's age of 15 months
  Improvements in maternal reports of positive emotional responses to their babies
Parental Acceptance (measured with the Parental Acceptance and Rejection Questionnaire) | Assessment at child's age of 15 months
  Improvements in maternal reports of acceptance in parent-child relationships

CONTACTS AND LOCATIONS:
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No